CLINICAL TRIAL: NCT02260505
Title: A Randomized Multicenter Phase III Trial Evaluating the Interest of Imatinib Treatment Maintenance or Interruption After 3 Years of Adjuvant Treatment in Patients With Gastrointestinal Stromal Tumours (GIST)
Brief Title: Efficiency of Imatinib Treatment Maintenance or Interruption After 3 Years of Adjuvant Treatment in Patients With Gastrointestinal Stromal Tumours (GIST)
Acronym: ImadGist
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMADGIST; 2013-001372-37 (EudraCT Number)
Record Dates: First submitted 2014-07-30; First posted 2014-10-09 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Stromal Tumors; Resected Gastrointestinal Stromal Tumors; Non-metastatic; High Risk of Recurrence; KIT Gene Mutation
Keywords: Gastrointestinal Stromal Tumors; Non-metastatic; KIT +; Imatinib; Adjuvant treatment; High risk of recurrence; Tyrosine kinase inhibitor; Disease Free Survival; Overall survival; Time To Secondary Resistance; Safety profile; Quality of Life during treatment
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib maintenance (Experimental): Maintenance of Imatinib at the last dose routinely taken by the patient in the 3 years period prior to randomization (either 300 or 400 mg/day). Increase dose up to 800 mg/day if relapse according to RECIST 1.1 criteria. Any relapse/progressive disease at 800 mg/day will lead to Imatinib permanent discontinuation and study discontinuation. In case of toxicity, Imatinib dose will be interrupted or adjusted in accordance with Imatinib Specific Product Characteristics (SPC).
  Interventions: Drug: Imatinib maintenance
- Imatinib Interruption (No Intervention): Treatment corresponding to standard practice : interruption of Imatinib from the day of randomization. Reintroduction of Imatinib at 400 mg/day after first relapse according to RECIST 1.1 criteria; Then increase dose to 800 mg/day after 2d relapse. Any relapse/progressive disease at 800 mg/day will lead to Imatinib permanent discontinuation and study discontinuation. In case of toxicity, Imatinib dose will be interrupted or adjusted in accordance with Imatinib SPC.

INTERVENTIONS:
Drug: Imatinib maintenance — Either 300 or 400 mg/day in accordance with the last dose routinely taken by the patient in the 3-year period before randomization. The treatment will be orally taken at time of meal with a large glass of water
  Other Names: Glivec; Imatinib mésilate
  Arms: Imatinib maintenance

SUMMARY:
This is a 2 arms study concerning patients with primary GIST who followed an Imatinib adjuvant treatment for 3 years after surgery and who have a high risk of recurrence.

In the first arm, patients will continue Imatinib treatment for 3 more years, allowing to determine if the continuation of this treatment is efficient for disease control, in terms of Disease Free Survival improvement.

In the second arm, patients will discontinue the Imatinib treatment, as standard practice. This arm will allow to determine if the re-introduction of Imatinib at relapse is still an efficient treatment for the control of disease.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumours (GISTs) are rare mesenchymal neoplasms, mostly diagnosed between 55 and 60 years of age, which account for 5% of all sarcomas. Worldwide annual incidence is approximately 12 cases per million people, corresponding to approximately 800 new cases per year in France.

A large majority of GISTs harbour activating mutations in the proto-oncogenes KIT and/or PDGFRA, both coding cell-surface cytokine receptors with tyrosine-protein kinase activity.

Imatinib mesilate (Glivec®, Novartis Pharma SAS) is a selective tyrosine kinase inhibitor, leading to inhibition of KIT and PDGFRA signalling pathways. The introduction of imatinib has revolutionised the therapeutic management of GIST patients and has provided an unprecedented demonstration of the clinical benefit of a targeted therapy for patients with advanced/metastatic solid tumors. First results from prospective trials conducted with imatinib in GIST patients have demonstrated a 300% increase in median overall survival, and a likely 100% increase in 5 and 10-year survival as compared to cytotoxic chemotherapy.

The successful use of imatinib in the treatment of advanced GISTs and the significant risk of recurrence of advanced GISTs have prompted the investigation of the clinical benefit of imatinib as a post-operative adjuvant therapy. Two prospective randomized Phase III trials have demonstrated that adjuvant imatinib treatment significantly prolong overall survival (OS) and recurrence-free survival (RFS) when given for 3 years. To date, imatinib is also indicated in the adjuvant setting after complete resection of primary, localized, KIT-positive GIST at high risk of recurrence. However, the optimal treatment duration remains unclear and it should be determined whether

1. prolonged use of adjuvant imatinib beyond 3 years may enable to reduce the risk of GIST recurrence and to improve overall survival, and
2. imatinib rechallenge is efficient for treating recurrence after completion of 3-year adjuvant imatinib therapy.

This trial is an open-label, randomized, multicenter phase III study aiming to determine the clinical impact of maintaining imatinib treatment beyond 3 years in the adjuvant setting for patients with resected GISTs at high risk of recurrence according to the National Comprehensive Cancer Network Task Force on GIST (NCCN) risk classification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study
* Patients must have histologically confirmed diagnosis of localized GIST with documented KIT (CD117) positivity (by polyclonal DAKO antibody staining)
* Documented macroscopically complete surgical R0 or R1 resection of primary GIST lesion with no evidence of residual lesions or metastases on the baseline CT-scan or MRI performed no more than 4 weeks before randomization.
* Risk of tumor recurrence ≥ 35% according to National Comprehensive Cancer Network Task Force on GIST (NCCN) risk classification (Demetri et al., 2010) (See Appendix 1)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients must be under imatinib treatment (at 300 or 400 mg/day) initiated immediately after resection and maintained for 3 years (i.e. 36 months ± 3 months at the time of randomization) with no more than 3 consecutive months or 6 months in total of interruption during these past 3 years.
* Patients must have normal organ and bone marrow function at baseline as defined below:

  * absolute neutrophil count (ANC) ≥ 1.5 G/L, platelet count ≥ 100 G/L, and haemoglobin of ≥ 9 g/dL).
  * Serum total bilirubin ≤ 1.5 (upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (or 5 x ULN in case of hepatic metastases at time of reintroduction)
  * Adequate renal function assessed by at least one of the following:

    * 1) Serum creatinine ≤ 1.5 x ULN or
    * 2) creatinine clearance estimate ≥ 50 mL/min (as calculated according to Cockcroft-Gault formula or MDRD formula for patients > 65 years).
* Recovered from prior anti-neoplasia treatment-related toxicity (persistent treatment-related toxicity < Grade 2 as per Common Toxicity Criteria for Adverse Effects (CTCAE) v4 are accepted)
* Women of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to randomization. A positive urine test must be confirmed by a serum pregnancy test
* Patient must use effective contraception at least 4 weeks prior to study entry, during the study participation and for at least 30 days post-treatment (not applicable for women of non-childbearing potential)
* Ability to understand and willingness for follow-up visits.
* Covered by a medical insurance.
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient concurrently using other approved or investigational antineoplastic agents
* Any contra-indication to imatinib treatment as per Glivec® SPC
* Patient with GIST harboring the mutation D842V in PDGFRA
* Major concurrent disease affecting cardiovascular system, liver, kidneys, haematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures or results.
* Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years.
* Patient receiving concurrent treatment with warfarin (acceptable alternative: low-molecular weight heparin) or any prohibited concomitant and/or concurrent medications
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Major surgery within 2 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 6 years (i.e. at the the time of last patient last visit)
  Time from the date of randomisation to the first documented relapse or death due to any cause. Patients with no event at the time of analysis will be censored at the date of the last adequate tumour assessment. The results will be analyzed according to the study arm and randomization strata to wich patients were assigned.

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 years (i.e. at the the time of last patient last visit)
  Time from the date of randomization until the date of death due to any cause and censored at the date of last contact for patients alive at last contact. The results will be analyzed according to the study arm and randomization strata to wich patients were assigned.
Time to Secondary Resistance (TSR) | 6 years (i.e. at the the time of last patient last visit)
  Time from the date of randomization until the date of first relapse under Imatinib treatment (i.e first relapse in the "Imatinib maintenance arm" and relapse after reintroduction of Imatinib in the "Interruption of Imatinib arm"). The results will be analyzed according to the study arm and randomization strata to wich patients were assigned.
Percentage of patients in Complete Response (%CR) in interruption arm after reintroduction of Imatinib | 6 years (i.e. at the the time of last patient last visit)
  Percentage of patients in Complete Response (CR) after reintroduction of Imatinib treatment for patients assigned to the interruption arm and who experience GIST recurrence. CR is assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Frequency of Adverse Events (AE) | 6 years (i.e. at the the time of last patient last visit)
  The assessment of safety will be based mainly on the frequency of AE based on the Common Toxicity Criteria version 4 grade. AE will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Descriptive statistics will be provided for characterizing and assessing patient tolerance to treatment. Patients with at least either one serious AE, or one grade 3-4, or one AE requiring the interruption of study treatment, will be described by study arm and compared using a Pearson's Chi2 test or a Fisher's exact test, if adequate. Patients will be analyzed according the duration of exposure to imatinib
Patient's Quality of Life (QoL) | 6 years (i.e at the the time of last patient last visit)
  QoL will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire (QLQ-C30). Descriptive statistics (e.g. means and medians) will be used to summarize the scored scales at it scheduled assessment time point of the questionnaire. The distribution of time to definitive health-related QoL deterioration by study arms will be estimated using the Kaplan-Meier method. The time to definitive deterioration is defined as the time from the date of randomization to the date of event, wich is defined as > 10 points decrease from baseline of QLQ-C30 global score (items 29 and 30) or death due to any cause. If patient has not had an event, time to QoL deterioration will be censored at the date of last adequate evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, Pr, Principal Investigator — Centre Léon Bérard, Lyon
Locations (17):
- France (17):
  - Institut Paoli-Calmettes, Marseille, Bouches Du Rhône
  - Centre Hospitalier Universitaire La Timone, Marseille, Bouches Du Rhône
  - Centre Georges François Leclerc, Dijon, Côte d'Or
  - CHRU de Besançon - Hôpital Minjoz, Besançon, Doubs
  - Institut Bergonié, Bordeaux, Gironde
  - Centre Régional de Lutte contre le Cancer de Montpellier, Montpellier, Hérault
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire Atlantique
  - Centre Hospitalier universitaire Robert Debré, Reims, Marne
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Centre Oscar Lambret, Lille, Nord
  - Institut de cancérologie LUCIEN NEUWIRTH, Saint-priest-en-jarez, Pays de la Loire Region
  - Centre Léon Bérard, Lyon, Rhône
  - Institut de Cancérologie Gustave Roussy, Villejuif, Val De Marne
  - AP-HP Hôpital Saint-Antoine, Paris
  - Centre Eugène Marquis, Rennes
  - CHRU Strasbourg - Hôpital Hautepierre, Strasbourg
  - AP-HP Hôpital Européen Georges Pompidou, Paris, Île-de-France Region

REFERENCES:
- [Background] Blackstein ME, Blay JY, Corless C, Driman DK, Riddell R, Soulieres D, Swallow CJ, Verma S; Canadian Advisory Committee on GIST. Gastrointestinal stromal tumours: consensus statement on diagnosis and treatment. Can J Gastroenterol. 2006 Mar;20(3):157-63. doi: 10.1155/2006/434761. PMID 16550259
- [Background] Blanke CD, Demetri GD, von Mehren M, Heinrich MC, Eisenberg B, Fletcher JA, Corless CL, Fletcher CD, Roberts PJ, Heinz D, Wehre E, Nikolova Z, Joensuu H. Long-term results from a randomized phase II trial of standard- versus higher-dose imatinib mesylate for patients with unresectable or metastatic gastrointestinal stromal tumors expressing KIT. J Clin Oncol. 2008 Feb 1;26(4):620-5. doi: 10.1200/JCO.2007.13.4403. PMID 18235121
- [Background] Blanke CD, Rankin C, Demetri GD, Ryan CW, von Mehren M, Benjamin RS, Raymond AK, Bramwell VH, Baker LH, Maki RG, Tanaka M, Hecht JR, Heinrich MC, Fletcher CD, Crowley JJ, Borden EC. Phase III randomized, intergroup trial assessing imatinib mesylate at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumors expressing the kit receptor tyrosine kinase: S0033. J Clin Oncol. 2008 Feb 1;26(4):626-32. doi: 10.1200/JCO.2007.13.4452. PMID 18235122
- [Background] Blay JY, von Mehren M, Blackstein ME. Perspective on updated treatment guidelines for patients with gastrointestinal stromal tumors. Cancer. 2010 Nov 15;116(22):5126-37. doi: 10.1002/cncr.25267. PMID 20661913
- [Background] Blay JY, Le Cesne A, Ray-Coquard I, Bui B, Duffaud F, Delbaldo C, Adenis A, Viens P, Rios M, Bompas E, Cupissol D, Guillemet C, Kerbrat P, Fayette J, Chabaud S, Berthaud P, Perol D. Prospective multicentric randomized phase III study of imatinib in patients with advanced gastrointestinal stromal tumors comparing interruption versus continuation of treatment beyond 1 year: the French Sarcoma Group. J Clin Oncol. 2007 Mar 20;25(9):1107-13. doi: 10.1200/JCO.2006.09.0183. PMID 17369574
- [Background] Casali PG, Jost L, Reichardt P, Schlemmer M, Blay JY; ESMO Guidelines Working Group. Gastrointestinal stromal tumors: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2008 May;19 Suppl 2:ii35-8. doi: 10.1093/annonc/mdn080. No abstract available. PMID 18456761
- [Background] ClinicalTrials.gov. Imatinib mesilate or observation only in treating patients who have undergone surgery for localized gastrointestinal stromal tumor. NCT identifier: NCT00103168. 13-12-2009. Ref Type: Online Source
- [Background] ClinicalTrials.gov. Five year adjuvant imatinib mesilate (Gleevec®) in gastrointestinal stromal tumor (GIST). NCT Identifier: NCT00867113. 24-8-2011. Ref Type: Online Source
- [Background] Corless CL, Heinrich MC. Molecular pathobiology of gastrointestinal stromal sarcomas. Annu Rev Pathol. 2008;3:557-86. doi: 10.1146/annurev.pathmechdis.3.121806.151538. PMID 18039140
- [Background] Corless CL, Barnett CM, Heinrich MC. Gastrointestinal stromal tumours: origin and molecular oncology. Nat Rev Cancer. 2011 Nov 17;11(12):865-78. doi: 10.1038/nrc3143. PMID 22089421
- [Background] Dematteo RP, Ballman KV, Antonescu CR, Maki RG, Pisters PW, Demetri GD, Blackstein ME, Blanke CD, von Mehren M, Brennan MF, Patel S, McCarter MD, Polikoff JA, Tan BR, Owzar K; American College of Surgeons Oncology Group (ACOSOG) Intergroup Adjuvant GIST Study Team. Adjuvant imatinib mesylate after resection of localised, primary gastrointestinal stromal tumour: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Mar 28;373(9669):1097-104. doi: 10.1016/S0140-6736(09)60500-6. Epub 2009 Mar 18. PMID 19303137
- [Background] DeMatteo RP, Lewis JJ, Leung D, Mudan SS, Woodruff JM, Brennan MF. Two hundred gastrointestinal stromal tumors: recurrence patterns and prognostic factors for survival. Ann Surg. 2000 Jan;231(1):51-8. doi: 10.1097/00000658-200001000-00008. PMID 10636102
- [Background] Dematteo RP, Heinrich MC, El-Rifai WM, Demetri G. Clinical management of gastrointestinal stromal tumors: before and after STI-571. Hum Pathol. 2002 May;33(5):466-77. doi: 10.1053/hupa.2002.124122. PMID 12094371
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Background] Patrikidou A, Chabaud S, Ray-Coquard I, Bui BN, Adenis A, Rios M, Bertucci F, Duffaud F, Chevreau C, Cupissol D, Domont J, Perol D, Blay JY, Le Cesne A; French Sarcoma Group. Influence of imatinib interruption and rechallenge on the residual disease in patients with advanced GIST: results of the BFR14 prospective French Sarcoma Group randomised, phase III trial. Ann Oncol. 2013 Apr;24(4):1087-93. doi: 10.1093/annonc/mds587. Epub 2012 Nov 21. PMID 23175622
- [Background] Gold JS, Gonen M, Gutierrez A, Broto JM, Garcia-del-Muro X, Smyrk TC, Maki RG, Singer S, Brennan MF, Antonescu CR, Donohue JH, DeMatteo RP. Development and validation of a prognostic nomogram for recurrence-free survival after complete surgical resection of localised primary gastrointestinal stromal tumour: a retrospective analysis. Lancet Oncol. 2009 Nov;10(11):1045-52. doi: 10.1016/S1470-2045(09)70242-6. Epub 2009 Sep 28. PMID 19793678
- [Background] H.Joensuu, M.Eriksson, J.Hatrmann, K.Sundby Hall, J.Schutte, A. Reichardt, M.Schlemmer, E. Wardelmann, G.Ramadori, S. E. Al-Batran B. E. Nilsson O. Monge R. Kallio, and M.Sarlomo-Rikala, P. Bono M. Leinonen P. Hohenberger T. Alvegard P. Reichardt. Three years of imatinib improves survival for high-risk gastrointestinal stromal tumours. ASCO 2011 . 2011. Ref Type: Abstract
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Hirota S, Isozaki K, Moriyama Y, Hashimoto K, Nishida T, Ishiguro S, Kawano K, Hanada M, Kurata A, Takeda M, Muhammad Tunio G, Matsuzawa Y, Kanakura Y, Shinomura Y, Kitamura Y. Gain-of-function mutations of c-kit in human gastrointestinal stromal tumors. Science. 1998 Jan 23;279(5350):577-80. doi: 10.1126/science.279.5350.577. PMID 9438854
- [Background] Jiang WZ, Guan GX, Lu HS, Yang YH, Kang DY, Huang HG. Adjuvant imatinib treatment after R0 resection for patients with high-risk gastrointestinal stromal tumors: a median follow-up of 44 months. J Surg Oncol. 2011 Dec;104(7):760-4. doi: 10.1002/jso.22010. Epub 2011 Jun 28. PMID 21713778
- [Background] Joensuu,H. and Ericksson,M.H.J. (2011). Twelve versus 36 monts of adjuvant imatinib as treatment of operable GIST with high risk of recurrence: Final results of a randomized trial (SSGXVIII/AIO). J. Clin. Oncol.
- [Background] Joensuu H, Vehtari A, Riihimaki J, Nishida T, Steigen SE, Brabec P, Plank L, Nilsson B, Cirilli C, Braconi C, Bordoni A, Magnusson MK, Linke Z, Sufliarsky J, Federico M, Jonasson JG, Dei Tos AP, Rutkowski P. Risk of recurrence of gastrointestinal stromal tumour after surgery: an analysis of pooled population-based cohorts. Lancet Oncol. 2012 Mar;13(3):265-74. doi: 10.1016/S1470-2045(11)70299-6. Epub 2011 Dec 6. PMID 22153892
- [Background] Le Cesne,A., Ray-Coquard,I.L., Bui Nguyen,B., Adenis,A., Rios,M., Bertucci,F., Duffaud,F., Cupissol,D., Chevreau,C., Bompas,E., Cioffi,A., Chabaud,S., Perol,D., and Blay,J. (2011). Time to secondary resistance (TSR) after interruption of imatinib (IM) in advanced GIST: Updated results of the prospective French Sarcoma Group randomized phase III trial on long-term survival. ASCO Meeting Abstracts 29, 10015.
- [Background] Le Cesne A, Ray-Coquard I, Bui BN, Adenis A, Rios M, Bertucci F, Duffaud F, Chevreau C, Cupissol D, Cioffi A, Emile JF, Chabaud S, Perol D, Blay JY; French Sarcoma Group. Discontinuation of imatinib in patients with advanced gastrointestinal stromal tumours after 3 years of treatment: an open-label multicentre randomised phase 3 trial. Lancet Oncol. 2010 Oct;11(10):942-9. doi: 10.1016/S1470-2045(10)70222-9. Epub 2010 Sep 21. PMID 20864406
- [Background] Pisters PW, Colombo C. Adjuvant imatinib therapy for gastrointestinal stromal tumors. J Surg Oncol. 2011 Dec;104(8):896-900. doi: 10.1002/jso.22002. PMID 22069174
- [Background] Ray-Coquard,I.L., Bin Bui,N., Adenis,A., Rios,M., Bertucci,F., Chabaud,S., Perol,D., Blay,J., Le Cesne,A., and Groupe Sarcome Francais & Groupe d'Etude des Tumeurs Osseuses (GSF-GETO) (2010). Risk of relapse with imatinib (IM) discontinuation at 5 years in advanced GIST patients: Results of the prospective BFR14 randomized phase III study comparing interruption versus continuation of IM at 5 years of treatment: A French Sarcoma Group Study. ASCO Meeting Abstracts 28, 10032.
- [Background] Tryggvason G, Gislason HG, Magnusson MK, Jonasson JG. Gastrointestinal stromal tumors in Iceland, 1990-2003: the icelandic GIST study, a population-based incidence and pathologic risk stratification study. Int J Cancer. 2005 Nov 1;117(2):289-93. doi: 10.1002/ijc.21167. PMID 15900576
- [Background] Tzen CY, Wang JH, Huang YJ, Wang MN, Lin PC, Lai GL, Wu CY, Tzen CY. Incidence of gastrointestinal stromal tumor: a retrospective study based on immunohistochemical and mutational analyses. Dig Dis Sci. 2007 Mar;52(3):792-7. doi: 10.1007/s10620-006-9480-y. PMID 17253141
- [Background] Verweij J, Casali PG, Zalcberg J, LeCesne A, Reichardt P, Blay JY, Issels R, van Oosterom A, Hogendoorn PC, Van Glabbeke M, Bertulli R, Judson I. Progression-free survival in gastrointestinal stromal tumours with high-dose imatinib: randomised trial. Lancet. 2004 Sep 25-Oct 1;364(9440):1127-34. doi: 10.1016/S0140-6736(04)17098-0. PMID 15451219